CLINICAL TRIAL: NCT00637091
Title: A Phase II Trial of Cetuximab Plus Irinotecan as a 2nd-line Treatment in Patients With Metastatic Colorectal Cancer After Failure to Irinotecan That Express Wild-type KRAS With and Without Detectable EGFR Expression
Brief Title: Efficacy Analysis of Cetuximab Plus Irinotecan in Patients With Wild-type KRAS Without Regard to Epidermal Growth Factor Receptor (EGFR) Expressions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Tae Won Kim, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC-ONCGI-2008-0031
Record Dates: First submitted 2008-03-10; First posted 2008-03-17 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Advanced Colorectal Cancer
MeSH Terms: interventions — Cetuximab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EGFR expression (Experimental): Patients' accrual will be adjusted by EGFR expression (positive vs. negative)
  Interventions: Drug: Cetuximab, irinotecan

INTERVENTIONS:
Drug: Cetuximab, irinotecan — cetuximab, irinotecan
  Other Names: PharmDx kit for EGFR staining.

SUMMARY:
The purpose of this study is to investigate the response rate of cetuximab plus irinotecan every 2 weeks in patients harboring wild-type KRAS with and without detectable EGFR-expressing metastatic CRC after failure to irinotecan in an exploratory manner.

DETAILED DESCRIPTION:
Twenty patients with positive-EGFR results and 20 patients with negative-EGFR results will be accrued in this study. All patients should have wild-type KRAS.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal adenocarcinoma, Wild KRAS, 18-75 yr
* Estimated life expectancy of more than 3 months
* ECOG performance status of 0 to 1 at study entry
* Adequate bone marrow function
* Adequate liver function
* Documented progression during or within 3 months of irinotecan-containing regimens as a first-line chemotherapy
* Immunohistochemical evidence of a presence or absence of EGFR expression by PharmDx Kit
* Informed Consent

Exclusion Criteria:

* Central nervous system (CNS) metastases or prior radiation for CNS metastases.
* Intestinal obstruction or impending intestinal obstruction due to peritoneal carcinomatosis
* Surgery (excluding biopsy for diagnosis) during 4 weeks prior to inclusion in the study.
* Evidence of gastrointestinal bleeding
* Exposure to Cetuximab
* Prior administration of monoclonal antibodies, EGFR signal transduction inhibitors or EGFR-targeted treatment
* KRAS mutant Status
* Patients with serious toxicity to previous irinotecan-based chemotherapy
* Other serious illness or medical conditions

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-03; Primary Completion 2009-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Response rate | 8 week

SECONDARY OUTCOMES:
Progression free survival, overall survival | every 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Result] Kang MJ, Hong YS, Kim KP, Kim SY, Baek JY, Ryu MH, Lee JL, Chang HM, Kim MJ, Chang HJ, Kang YK, Kim TW. Biweekly cetuximab plus irinotecan as second-line chemotherapy for patients with irinotecan-refractory and KRAS wild-type metastatic colorectal cancer according to epidermal growth factor receptor expression status. Invest New Drugs. 2012 Aug;30(4):1607-13. doi: 10.1007/s10637-011-9703-8. Epub 2011 Jun 25. PMID 21706149